CLINICAL TRIAL: NCT06591767
Title: Potential Pharmacological Effects of Supplemental Quercetin in the Management of Mild to Moderate Hyperuricemia
Brief Title: Quercetin as Possible Supportive Therapy for Mild to Moderate Hyperuricemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: University of Urbino "Carlo Bo" (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 88_18.01.2023_QuercetinFit
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quercetin group (Experimental): In this group hyperuricemic patients (uric acid > 8 mg/dL) received oral supplemental Quercetin, twice a day for 90 days.
  Interventions: Dietary Supplement: Quercetin
- Control group 1 (Active Comparator): In this group hyperuricemic patients (uric acid > 8 mg/dL) received oral supplemental Berberine and monacolins based supplement, twice a day for 90 days.
  Interventions: Combination Product: Berberol K®
- Control group 2 (Active Comparator): In this group normouricemic patients (uric acid < 7 mg/dL) received oral supplemental Berberine and monacolins based supplement, twice a day for 90 days.
  Interventions: Combination Product: Berberol K®

INTERVENTIONS:
Dietary Supplement: Quercetin — 200 mg supplemental Quercefit®
  Other Names: Quevir®
  Arms: Quercetin group
Combination Product: Berberol K® — Berberine Phytosome® 730 mg
  + MonakoPure® containing 2.9 mg of monacolin K and KA from red yeast rice extract
  Arms: Control group 1; Control group 2

SUMMARY:
Uric acid, a metabolic byproduct of purine degradation in humans, is a known risk factor for conditions such as gout and type 2 diabetes. Research has shown that supplementation with quercetin can significantly reduce plasma uric acid levels in individuals with mild hyperuricemia, potentially mitigating these associated risks.

DETAILED DESCRIPTION:
Uric acid, a metabolic byproduct of purine degradation in humans, is a significant risk factor for the development of gout and type 2 diabetes. Supplementation with quercetin, a flavonol not naturally produced by the human body, has been shown to significantly reduce plasma uric acid levels in individuals with mild hyperuricemia. This effect is primarily achieved through the inhibition of xanthine oxidoreductase, an enzyme crucial to uric acid production.

Quercetin is the most abundant polyphenol found in fruits and vegetables and is widely used as a dietary supplement to boost the immune system and promote overall health. It is characterized by three key properties: antioxidant, anti-inflammatory, and immunomodulatory. These combined actions make quercetin a promising candidate for supporting various health conditions where oxidative stress, inflammation, and immune function play a role, including cardiovascular health, healthy aging, bone and joint health, sports and physical activity, gut health, and respiratory well-being.

The above-described properties of quercetin prompted investigators to explore its potential uricosuric therapeutic effect in two clinical studies. The first study will assess this effect in a retrospective cohort of COVID-19 patients who received quercetin as a supplemental therapy. In the second study, its potential uricosuric therapeutic effect will be assessed in a randomized controlled prospective clinical trial involving patients with mild to moderate hyperuricemia.

ELIGIBILITY:
Inclusion criteria:

* Aged between 18 and 75 years.
* Diagnosed with obesity.
* Diagnosed with hypercholesterolemia.
* With or without moderate hyperuricemia (serum uric acid ≥ 8 mg/dL).
* No restrictions on BMI, alcohol consumption, or smoking habits.

Exclusion criteria:

* Current use of uric acid-lowering medications (e.g., allopurinol, febuxostat).
* Diagnosed with oncological diseases.
* Diagnosed with neurological diseases.
* Diagnosed with inflammatory bowel diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Effect on circulatory uric acid | 90 days
  Change in plasma uric acid level

SECONDARY OUTCOMES:
Effect on lipids | 90 days
  Change in plasma cholesterol level
Effect on lipids | 90 days
  Change in plasma triglycerides level
Effect on glycemia | 90 days
  Change in plasma glucose level
Effect on glycemia | 90 days
  Change in plasma insulin level
Effect on body internal organs muscles | 90 days
  Change in the Creatine Phosphokinase (CPK) levels
Effect on liver function | 90 days
  Change in the Alanine Aminotransferase levels
Effect on liver function | 90 days
  Change in the Aspartate Aminotransferase levels
Effect on liver function | 90 days
  Change in the Alkaline Phosphatase levels
Effect on liver function | 90 days
  Change in the Gamma-Glutamyl Transferase levels
Effect on liver function | 90 days
  Change in the Bilirubin levels
Supplement safety and tolerability | 90 days
  Number of patients reporting possible side effects

CONTACTS AND LOCATIONS:
Locations (1):
- S. Orsola-Malpighi Polyclinic Hospital, Bologna, Italy